CLINICAL TRIAL: NCT05346536
Title: Liquid Biopsy and Pancreas Cancer: Detection of AXL(+) Functional CTCs Using EPIDROP
Brief Title: Liquid Biopsy and Pancreas Cancer: Detection of AXL(+) CTCs (CTC-AXL-PANC)
Acronym: CTC-AXL-PANC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0024
Record Dates: First submitted 2022-04-19; First posted 2022-04-26 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Cancer; Circulating Tumor Cell
Keywords: Metastatic Pancreatic Cancer; Circulating Tumor Cell; AXL; CellSearch
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Intervention Model Description: Single-centre prospective cohort Cohort of newly diagnosed major patients with metastatic pancreatic cancer, naïve of any treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metastatic pancreatic cancer treatment-naive patients (Experimental): Newly diagnosed major patients with metastatic pancreatic cancer, naïve of any treatment for metastatic disease
  Interventions: Other: Detection of circulating tumor cells expressing Axl: CTC-AXL(+)

INTERVENTIONS:
Other: Detection of circulating tumor cells expressing Axl: CTC-AXL(+) — Detection of CTC-AXL(+) using 2 techniques:
  * CellSearch®, FDA-USA approved technology
  * EPIDROP System
  CellSearch® (Menarini Company) The current gold-standard CellSearch® technique requires the use of CellSave tubes. This technique allows the isolation of fixed CTCs. This technique uses a positive (CellSearch® Epithelial Cell Kit) enrichment method from total blood using magnetic beads coupled to an EpCAM capture antibody. CTCs are then detected (anti-panCK antibodies, DAPI, anti-CD45 and characterized (anti-AXL antibody) by immunofluorescence (IF).
  EPIDROP It requires the use of EDTA tubes. This technique is based on a method of negative enrichment of CTCs from total blood using a cocktail of tetrameric antibodies to eliminate unwanted blood cells and to preserve only purified tumor cells (RosetteSep - StemCell Technology).Then, cells are loaded in a microfluidic chip. The detection and characterization is done by IF to the single cell in micro-droplets.

SUMMARY:
In solid cancers, some more aggressive tumor cells actively detach from the primary lesion and then travel through the circulating compartment to reach distant organs and form micro-metastases. These circulating tumor cells (CTCs) that have become disseminated tumor cells (DTCs) flourish in their new environments and may remain dormant for many years after the complete resection of the primary tumor. Detecting CTCs in the blood is also relevant for assessing tumor progression, prognosis and therapeutic follow-up. The non-invasive, highly sensitive for CTCs analysis is called "liquid biopsy". Pancreatic adenocarcinoma and breast cancer remain among cancers of very poor prognosis and thus represent a major therapeutic challenge. In recent years, the Axl membrane tyrosine kinase receptor has been the target of growing interest. Activation of the Gas6/Axl signaling pathway is associated with, among other things, tumor cell growth and survival, epithelial to mesenchymal transition (EMT) or drug resistances. In addition, Axl overexpression is frequently identified in patients with pancreatic adenocarcinoma and is associated with a poor prognosis. For example, the Laboratoire des Cellules Circulantes Rares Humaines (LCCRH) at the CHU and the University of Montpellier has developed two new "CTC-AXL" tests to detect CTCs expressing Axl: one using the CellSearch® (gold standard and FDA-approved) system and the other using the EPIDROP technique. The purpose of this research project is to assess the concordance of the "CTC-AXL" measurement by the innovative EPIDROP technique and the CellSearch® technique in patients with metastatic pancreatic or breast cancer.

DETAILED DESCRIPTION:
In solid cancers, after the formation and growth of the primary tumor, some more aggressive tumor cells actively detach from it and then travel through the circulating compartment to reach distant organs (bone marrow - liver - lung - brain…) and constitute new foci or micro-metastases. These circulating tumor cells (CTCs) that have become disseminated tumor cells (DTCs) flourish in their new environments and may remain dormant for many years after the complete resection of the primary tumor. Due to events not fully elucidated, DTCs can develop on site giving rise to macroscopic metastases but also join again the circulating compartment in the form of CTCs, swarm, colonize other organs and cause secondary metastases.

Detecting CTCs in the blood is very relevant for assessing tumor progression but also promising in terms of cancer disease prognosis and therapeutic follow-up. This new approach, published for the first time in 2010 under the term liquid biopsy, is therefore defined as a non-invasive blood test, extremely sensitive, achievable in real time and that allows the analysis of CTCs.

Currently, the choice of targeted therapies for a given patient is made after analyzing the primary tumor for expression and/or genomic status of specific molecular targets.

Many studies show that metastatic cells have phenotypic and genotypic characteristics distinct from those of most of the primary tumor. This can be explained either because metastatic cells acquire new genomic skills over time, or because a subset of metastatic sub-clone pre-exists within the primary tumor but has escaped detection by standard tissue biopsy techniques.

A direct analysis of CTCs could provide important additional information to prevent patients from inappropriate, costly treatments and harmful side effects.

For several years, the AXL protein, a tyrosine kinase receptor, has emerged as a new strategic target in oncology. Over-expression of AXL has been frequently identified in patients with pancreatic adenocarcinoma. AXL is a member of the Tyro3-Axl-Mer family, like its ligand protein Gas-6 (growth arrest-specific). An activation of the Gas6/AXL signaling pathway results in the activation of several effector pathways such as RAS/RAF/MEK/ERK or PI3K/AKT and is associated with, among other things, tumor cell growth and survival, metastatic formation and dissemination, Epithelial-to-mesenchymal transition (EMT) or drug resistances. It has been shown clinically that the AXL protein is a factor of poor prognosis and resistance to reference treatments (radiotherapy, chemotherapy or targeted therapy). Thus, many therapeutic strategies have been proposed and developed to inhibit the AXL pathway, ranging from chemical molecules, blocking its kinase activity and therefore the underlying signaling pathways, to nucleotide aptamers, AXL fusion proteins, and monoclonal antibodies.

Pancreatic adenocarcinoma, the 4th leading of cancer related deaths, remains among cancers of very poor prognosis and thus represents a major therapeutic challenge. The median overall survival is 11.1 months after optimal treatment (FOLFIRINOX). The clinical relevance and oncogenic potential of AXL in the progression of different types of tumors have been largely evidenced. Indeed, 50% to 75% of pancreatic adenocarcinoma samples have overexpression of AXL and the level of expression of AXL is correlated with clinical parameters indicating tumor aggressiveness and poor prognosis such as frequency of distant metastases or the survival.

In this context, the LCCRH lab, which has specialized in the detection and analysis of CTCs for 20 years, has developed a CTC-AXL detection test using the CellSearch® system. The CellSearch® system is the only method approved by the Food and Drug Administration (FDA) for the detection of CTC in colorectal, breast and metastatic prostate cancers. In addition, the LCCRH holds a patent for another technology for the detection and characterization of live and functional CTCs, called EPIDROP. The implementation of the AXL research is already done for AXL labelling on CTCs in EPIDROP as well as the visualization of the AXL cleavage by live CTC.

Thanks to this unique functional test of CTCs, it is easy to imagine offering an oncology 'oncogram' by testing in real time the effectiveness of drugs on CTCs and personalized medicine to patients.

This real-time liquid biopsy proposal on functional CTCs is quite innovative in Oncology.

To date, there are no studies on the study of functional CTCs related to AXL.

Primary objective:

- Evaluate the concordance of the CTC-AXL measurement (inclusive) by the innovative EPIDROP technique and the CellSearch technique®

Secondary objectives:

* Evaluate the accuracy of the CTC-AXL measurement (inclusive) between EPIDROP and CellSearch®
* Assess the degree of agreement between CTC-AXL measurement (inclusive) by EPIDROP and CellSearch®
* Evaluate the overall survival of patients with metastatic pancreatic cancer based on the number of circulating tumour cells carrying the AXL marker measured by EPIDROP or CellSearch® at inclusion
* Evaluate the progression-free survival of patients with metastatic pancreatic cancer based on the number of circulating tumour cells carrying the AXL marker measured by EPIDROP or CellSearch® at inclusion
* Culture CTCs from the blood sample (EDTA 10mL)
* Creation of a single liquid biopsy bio-bank for pancreatic cancer involving only plasma storage

  * Study the expression of PD-L1 (at inclusion) and detect the CTC subgroup expressing PD-L1 using EPIDROP and CellSearch® techniques;
  * Study the circulating immune system in this cohort of patients with metastatic pancreatic cancer by performing immunological analysis on blood mononuclear cells;
  * Determine if there is a significant correlation between the detection of CTC and CTC-PD-L1 and the circulating immune system (T cells, NK cells, B cells, macrophages, immune checkpoints, platelets);
  * To assess the correlation between CTC, CTC-PD-L1 and immune cells and the clinical outcomes (progression-free survival, overall survival) of these patients with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years old;
* Patients with pancreatic cancer with remote metastases, naïve of any treatment, that is, eligible for a first line of treatment;
* Patients with oral consent

Exclusion Criteria:

* Non-affiliation or non-beneficiary of a Social Security regimen;
* Frailty persons according to Article L1121-6 of the CSP;
* Adult protected or unable to give consent as per Article L1121-8 of the CPMP;
* Pregnant or lactating women as per MSC L1121-5.
* Not included for monitoring difficulties (mutation, insufficient motivation, predictable poor compliance, priority associated pathology in care, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
CTC-AXL measurement concordance rate | 30 days
  CTC-AXL measurement concordance rate by EPIDROP (AXL(-): 0 vs AXL(+): 1) and CellSearch® (AXL(-): 0 vs AXL(+): 1)

SECONDARY OUTCOMES:
Sensitivity (Se) defined as the proportion of AXL(+) positive patients (assessed by reference technique: CellSearch®) with a positive EPIDROP result | 30 days
Specificity (Sp) defined as the proportion of AXL(-) negative patients (assessed by reference technique: CellSearch®) with a negative result by EPIDROP | 30 days
Positive predictive value (PPV) defined as the proportion of patients with a positive EPIDROP result that is actually positive (as assessed by the reference technique: CellSearch®). | 30 days
Negative Predictive Value (VPN) defined as the proportion of patients, whose EPIDROP result is negative, that is effectively negative (assessed by reference technique: CellSearch®) | 30 days
Number of CTC-AXL at inclusion (0 vs 1 vs 2-3 vs 4 vs 5) measured by EPIDROP | 30 days
Number of CTC-AXL at inclusion (0 vs 1 vs 2-3 vs 4 vs 5) measured by the CellSearch technique® | 30 days
Overall Survival | 36 months
  Overall survival defined by the time between the date of diagnosis of the metastatic disease and the date of death regardless of the cause
Progression-Free Survival | 36 months
  Progression-free survival defined by the time between the date of diagnosis of the metastatic disease and the date of the 1st progression or the date of death regardless of the cause
Number of CTC at inclusion (0 vs 1 vs 2-3 vs 4 vs 5) measured by EPIDROP® | 30 days
Number of CTC at inclusion (0 vs 1 vs 2-3 vs 4 vs 5) measured by the CellSearch technique® | 30 days
CTC-PD-L1 measurement at inclusion (PD-L1(-): 0 vs PD-L1 (+): 1) measured by EPIDROP® | 30 days
CTC-PD-L1 measurement at inclusion (PD-L1(-): 0 vs PD-L1 (+): 1) measured by the CellSearch technique® | 30 days
Number of CTC-PD-L1 at inclusion (0 vs 1 vs 2-3 vs 4 vs 5) measured by EPIDROP® | 30 days
  Number of CTC labelled by anti-PD-L1 antibody detected by EPIDROP®
Number of CTC-PD-L1 at inclusion (0 vs 1 vs 2-3 vs 4 vs 5) measured by the CellSearch technique® | 30 days
  Number of CTC labelled by anti-PD-L1 antibody detected by CellSearch
Evaluation of circulating immune system: T cells | 30 days
Evaluation of circulating immune system: NK cells | 30 days
Evaluation of circulating immune system: B cells | 30 days
Evaluation of circulating immune system: macrophages | 30 days
Evaluation of circulating immune system: immune checkpoints | 30 days
Evaluation of circulating immune system: platelets | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Alix-Panabières, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pantel K, Alix-Panabieres C. Tumour microenvironment: informing on minimal residual disease in solid tumours. Nat Rev Clin Oncol. 2017 Jun;14(6):325-326. doi: 10.1038/nrclinonc.2017.53. Epub 2017 Apr 11. No abstract available. PMID 28397823
- [Background] Pantel K, Alix-Panabieres C. Liquid biopsy and minimal residual disease - latest advances and implications for cure. Nat Rev Clin Oncol. 2019 Jul;16(7):409-424. doi: 10.1038/s41571-019-0187-3. PMID 30796368
- [Background] Alix-Panabieres C. The future of liquid biopsy. Nature. 2020 Mar;579(7800):S9. doi: 10.1038/d41586-020-00844-5. No abstract available. PMID 32214259
- [Background] Pantel K, Alix-Panabieres C. Circulating tumour cells in cancer patients: challenges and perspectives. Trends Mol Med. 2010 Sep;16(9):398-406. doi: 10.1016/j.molmed.2010.07.001. Epub 2010 Jul 29. PMID 20667783
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Conroy T, Gavoille C, Adenis A. Metastatic pancreatic cancer: old drugs, new paradigms. Curr Opin Oncol. 2011 Jul;23(4):390-5. doi: 10.1097/CCO.0b013e3283473610. PMID 21505335
- [Background] Conroy T, Hammel P, Hebbar M, Ben Abdelghani M, Wei AC, Raoul JL, Chone L, Francois E, Artru P, Biagi JJ, Lecomte T, Assenat E, Faroux R, Ychou M, Volet J, Sauvanet A, Breysacher G, Di Fiore F, Cripps C, Kavan P, Texereau P, Bouhier-Leporrier K, Khemissa-Akouz F, Legoux JL, Juzyna B, Gourgou S, O'Callaghan CJ, Jouffroy-Zeller C, Rat P, Malka D, Castan F, Bachet JB; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. FOLFIRINOX or Gemcitabine as Adjuvant Therapy for Pancreatic Cancer. N Engl J Med. 2018 Dec 20;379(25):2395-2406. doi: 10.1056/NEJMoa1809775. PMID 30575490
- [Background] Sohal DPS, Kennedy EB, Cinar P, Conroy T, Copur MS, Crane CH, Garrido-Laguna I, Lau MW, Johnson T, Krishnamurthi S, Moravek C, O'Reilly EM, Philip PA, Pant S, Shah MA, Sahai V, Uronis HE, Zaidi N, Laheru D. Metastatic Pancreatic Cancer: ASCO Guideline Update. J Clin Oncol. 2020 Sep 20;38(27):3217-3230. doi: 10.1200/JCO.20.01364. Epub 2020 Aug 5. PMID 32755482
- [Background] Koorstra JB, Karikari CA, Feldmann G, Bisht S, Rojas PL, Offerhaus GJ, Alvarez H, Maitra A. The Axl receptor tyrosine kinase confers an adverse prognostic influence in pancreatic cancer and represents a new therapeutic target. Cancer Biol Ther. 2009 Apr;8(7):618-26. doi: 10.4161/cbt.8.7.7923. Epub 2009 Apr 22. PMID 19252414
- [Background] Leconet W, Larbouret C, Chardes T, Thomas G, Neiveyans M, Busson M, Jarlier M, Radosevic-Robin N, Pugniere M, Bernex F, Penault-Llorca F, Pasquet JM, Pelegrin A, Robert B. Preclinical validation of AXL receptor as a target for antibody-based pancreatic cancer immunotherapy. Oncogene. 2014 Nov 20;33(47):5405-14. doi: 10.1038/onc.2013.487. Epub 2013 Nov 18. PMID 24240689
- [Background] Kariolis MS, Miao YR, Jones DS 2nd, Kapur S, Mathews II, Giaccia AJ, Cochran JR. An engineered Axl 'decoy receptor' effectively silences the Gas6-Axl signaling axis. Nat Chem Biol. 2014 Nov;10(11):977-83. doi: 10.1038/nchembio.1636. Epub 2014 Sep 21. PMID 25242553
- [Background] Shen Y, Chen X, He J, Liao D, Zu X. Axl inhibitors as novel cancer therapeutic agents. Life Sci. 2018 Apr 1;198:99-111. doi: 10.1016/j.lfs.2018.02.033. Epub 2018 Feb 27. PMID 29496493
- [Background] Tai KY, Shieh YS, Lee CS, Shiah SG, Wu CW. Axl promotes cell invasion by inducing MMP-9 activity through activation of NF-kappaB and Brg-1. Oncogene. 2008 Jul 3;27(29):4044-55. doi: 10.1038/onc.2008.57. Epub 2008 Mar 17. PMID 18345028
- [Background] Li Y, Ye X, Tan C, Hongo JA, Zha J, Liu J, Kallop D, Ludlam MJ, Pei L. Axl as a potential therapeutic target in cancer: role of Axl in tumor growth, metastasis and angiogenesis. Oncogene. 2009 Oct 1;28(39):3442-55. doi: 10.1038/onc.2009.212. Epub 2009 Jul 27. PMID 19633687
- [Background] Antony J, Huang RY. AXL-Driven EMT State as a Targetable Conduit in Cancer. Cancer Res. 2017 Jul 15;77(14):3725-3732. doi: 10.1158/0008-5472.CAN-17-0392. Epub 2017 Jun 30. PMID 28667075
- [Background] Rankin EB, Fuh KC, Taylor TE, Krieg AJ, Musser M, Yuan J, Wei K, Kuo CJ, Longacre TA, Giaccia AJ. AXL is an essential factor and therapeutic target for metastatic ovarian cancer. Cancer Res. 2010 Oct 1;70(19):7570-9. doi: 10.1158/0008-5472.CAN-10-1267. Epub 2010 Sep 21. PMID 20858715
- [Background] Ye X, Li Y, Stawicki S, Couto S, Eastham-Anderson J, Kallop D, Weimer R, Wu Y, Pei L. An anti-Axl monoclonal antibody attenuates xenograft tumor growth and enhances the effect of multiple anticancer therapies. Oncogene. 2010 Sep 23;29(38):5254-64. doi: 10.1038/onc.2010.268. Epub 2010 Jul 5. PMID 20603615
- [Background] Cerchia L, Esposito CL, Camorani S, Rienzo A, Stasio L, Insabato L, Affuso A, de Franciscis V. Targeting Axl with an high-affinity inhibitory aptamer. Mol Ther. 2012 Dec;20(12):2291-303. doi: 10.1038/mt.2012.163. Epub 2012 Aug 21. PMID 22910292
- [Background] Wilson C, Ye X, Pham T, Lin E, Chan S, McNamara E, Neve RM, Belmont L, Koeppen H, Yauch RL, Ashkenazi A, Settleman J. AXL inhibition sensitizes mesenchymal cancer cells to antimitotic drugs. Cancer Res. 2014 Oct 15;74(20):5878-90. doi: 10.1158/0008-5472.CAN-14-1009. Epub 2014 Aug 14. PMID 25125659
- [Background] Feneyrolles C, Spenlinhauer A, Guiet L, Fauvel B, Dayde-Cazals B, Warnault P, Cheve G, Yasri A. Axl kinase as a key target for oncology: focus on small molecule inhibitors. Mol Cancer Ther. 2014 Sep;13(9):2141-8. doi: 10.1158/1535-7163.MCT-13-1083. Epub 2014 Aug 19. PMID 25139999
- [Background] Gjerdrum C, Tiron C, Hoiby T, Stefansson I, Haugen H, Sandal T, Collett K, Li S, McCormack E, Gjertsen BT, Micklem DR, Akslen LA, Glackin C, Lorens JB. Axl is an essential epithelial-to-mesenchymal transition-induced regulator of breast cancer metastasis and patient survival. Proc Natl Acad Sci U S A. 2010 Jan 19;107(3):1124-9. doi: 10.1073/pnas.0909333107. Epub 2009 Dec 28. PMID 20080645
- [Background] Song X, Wang H, Logsdon CD, Rashid A, Fleming JB, Abbruzzese JL, Gomez HF, Evans DB, Wang H. Overexpression of receptor tyrosine kinase Axl promotes tumor cell invasion and survival in pancreatic ductal adenocarcinoma. Cancer. 2011 Feb 15;117(4):734-43. doi: 10.1002/cncr.25483. Epub 2010 Oct 4. PMID 20922806
- [Background] Zhang S, Xu XS, Yang JX, Guo JH, Chao TF, Tong Y. The prognostic role of Gas6/Axl axis in solid malignancies: a meta-analysis and literature review. Onco Targets Ther. 2018 Jan 23;11:509-519. doi: 10.2147/OTT.S150952. eCollection 2018. PMID 29416351
- [Background] Yu W, Ge X, Lai X, Lv J, Wang Y. The up-regulation of Axl is associated with a poor prognosis and promotes proliferation in pancreatic ductal adenocarcinoma. Int J Clin Exp Pathol. 2019 May 1;12(5):1626-1633. eCollection 2019. PMID 31933980
- [Background] Jacot W, Mazel M, Mollevi C, Pouderoux S, D'Hondt V, Cayrefourcq L, Bourgier C, Boissiere-Michot F, Berrabah F, Lopez-Crapez E, Bidard FC, Viala M, Maudelonde T, Guiu S, Alix-Panabieres C. Clinical Correlations of Programmed Cell Death Ligand 1 Status in Liquid and Standard Biopsies in Breast Cancer. Clin Chem. 2020 Aug 1;66(8):1093-1101. doi: 10.1093/clinchem/hvaa121. PMID 32712650
- [Background] Sinoquet L, Jacot W, Gauthier L, Pouderoux S, Viala M, Cayrefourcq L, Quantin X, Alix-Panabieres C. Programmed Cell Death Ligand 1-Expressing Circulating Tumor Cells: A New Prognostic Biomarker in Non-Small Cell Lung Cancer. Clin Chem. 2021 Nov 1;67(11):1503-1512. doi: 10.1093/clinchem/hvab131. PMID 34355741
- [Background] Alix-Panabieres C, Pantel K. Liquid Biopsy: From Discovery to Clinical Application. Cancer Discov. 2021 Apr;11(4):858-873. doi: 10.1158/2159-8290.CD-20-1311. PMID 33811121